CLINICAL TRIAL: NCT04051606
Title: Regorafenib in Bevacizumab Refractory Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7318
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Regorafenib (Experimental): 160 mg regorafenib 3 weeks on/ one week off in participants with Avastin refractory Glioblastoma, continued until progression or toxicity. Participants will receive an MRI every 8 weeks.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib is a monotherapy during the study, oral administration at 160 mg once daily will be administered for 3 weeks on /1 week off.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of Regorafenib in patients with recurrent or progressive glioblastoma (GBM) who have progressed on bevacizumab. Regorafenib is FDA approved administered as monotherapy during the study.

22 total patients are expected to participate in this study. Even though a participant may meet all the criteria for participation, it is possible that they will not be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* The participant (or legally representative if applicable) provides written informed consent for the trial.
* Patients with histologically confirmed glioblastoma or other grade IV malignant glioma (i.e. gliosarcoma, small cell glioblastoma, etc.), recurrent after prior external-beam fractionated radiotherapy and temozolomide chemotherapy.
* Patients with documented radiographic progression following bevacizumab therapy for treatment of glioblastoma
* Patients with up to 3 prior recurrences are allowed (patients could have received bevacizumab or bevacizumab containing regimen either in first or second recurrence).
* Karnofsky performance status ≥ 70%.
* Patients must have the following laboratory values:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin (Hgb) > 9 g/dL
* Serum total bilirubin: ≤ 1.5 x ULN
* ALT and AST ≤ 3.0 x ULN
* Serum creatinine ≤ 1.5 x ULN
* Blood coagulation parameters: INR ≤ 1.5
* Minimum interval since completion of radiation treatment is 12 weeks
* Minimum interval since last drug therapy:
* 3 weeks since last non-cytotoxic therapy
* 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen
* 6 weeks since the completion of a nitrosourea containing chemotherapy regimen.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test. The definition of adequate contraception will be based on the judgment of the investigator.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least2 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast, adequately treated stage I or II cancer from which the patient is in complete remission. Patients with other prior malignancies must be disease-free for ≥ three years.
* Patients must be maintained on a stable or decreasing corticosteroid regimen from the time of their baseline scan until the start of treatment and/or for at least 5 days before starting treatment. The maximum dosing of corticosteroid therapy is 4mg/day.
* Life expectancy of at least 12 weeks (3 months).
* Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* Patients who have had previous treatment with Regorafenib
* Patients who have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury ≤ 4 weeks prior to starting study drug, or patients who have had minor procedures, percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury
* Patients with impaired cardiac function or clinically significant cardiac diseases, including any of the following:
* Congestive heart failure - New York Heart Association (NYHA) > Class II
* History or presence of serious uncontrolled ventricular arrhythmias. Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
* Clinically significant resting bradycardia (defined as bradycardia that required intervention)
* Active coronary artery disease defined as Any of the following within 6 months prior to starting study drug: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG)
* Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE) in the last 6 months
* Uncontrolled hypertension (defined by a SBP ≥ 160 mm Hg or DBP ≥ 100 mm Hg despite anti-hypertensive medications)
* Patients with cirrhosis, or active viral or nonviral hepatitis.
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol
* Pregnant or breast-feeding women
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human, chimeric, or humanized antibodies
* Patients with active bleeding or pathologic conditions that carry a high risk of bleeding, (i.e. hereditary hemorrhagic telangiectasia).
* Patients who are currently receiving anticoagulation treatment (warfarin is not allowed, low weight heparin is allowed). Evidence or history of bleeding diathesis or coagulopathy.
* Patients unwilling or unable to comply with the protocol
* Any hemorrhage or bleeding event ≥ NCI CTCAE v5.0 Grade 3 within 4 weeks prior to start of study medication.
* Patients with phaeochromocytoma.
* Ongoing infection > Grade 2 NCI-CTCAE v5.0.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Persistent proteinuria ≥ Grade 3 NCI-CTCAE v5.0 (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 5.0 Grade 2 dyspnea).
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.

Excluded therapies and medications, previous and concomitant

* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment (regorafenib, other agents being investigated in combination with regorafenib).
* Prior use of regorafenib.
* Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Therapeutic anticoagulation with Vitamin-K antagonists (e.g., warfarin)
* Use of any herbal remedy (e.g. St. John's wort [Hypericum perforatum]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Median overall survival (OS) | Up to 3 years from start of treatment
  Median overall survival (OS) in patients with recurrent or progressive GBM who have progressed on bevacizumab.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 3 years from start of treatment
  Safety and tolerability of regorafenib by CTCAE version 5.0. Safety and tolerability will be defined by the percent of participants experiencing >= grade 3 AE/SAE
Objective response rate (ORR) | Up to 3 years from start of treatment
  ORR by modified RANO criteria. ORR defined by modified RANO criteria . The percentage of patients that have at least 50% reduction in their tumor size in 2 dimensions.
Progression free survival at 6 months (PFS-6). | at 6 months from start of treatment
  Survival and absence of progressive disease at 6 months, with progression defined as >25% in the sum of products of the perpendicular diameters of CE lesions; evidence of new lesion(s).
Median time to progression (TTP) | Up to 3 years from start of treatment
  Time that takes a median patient to progress defined as >25% in the sum of products of the perpendicular diameters of CE lesions; evidence of new lesion(s).

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share main findings of the clinical study report (CSR)
Supporting Information: CSR